CLINICAL TRIAL: NCT07334132
Title: General Anaesthesia vs Spinal Anaesthesia: Patient Outcomes and Success in Outpatient Primary Total Knee and Hip Arthroplasty
Acronym: GASPS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Örebro University, Sweden (Other); Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASPS; 2024-520127-89-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-16; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Osteo Arthritis Knee and Hip; Osteo Arthritis; Inflammatory Joint Disease (IJD)
Keywords: Total Knee Arthroplasty; Total Hip Arthroplasty; Outpatient Surgery; Same-Day Discharge; Ambulatory Arthroplasty; General Anaesthesia; Spinal Anaesthesia; Neuraxial Anaesthesia; Total Intravenous Anaesthesia; Postoperative Recovery; Quality of Recovery; QoR-15; Postoperative Pain; Postoperative Nausea and Vomiting; PONV; Patient-Reported Outcomes; Health Economic Evaluation; Cost-Effectiveness; Randomized Clinical Trial
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Anesthesia, General; Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Masking Description: This trial uses a partial blinding strategy to minimise bias while accommodating the practical requirements of the interventions. Participants and clinical staff involved in preoperative care will be blinded to the assigned anaesthesia method until a few hours prior to surgery.
  The anaesthesia team responsible for administering the allocated intervention will not be blinded, as they must deliver the specific anaesthetic technique (GA or SA). Outcome assessors will not be blinded, as their interactions with participants and the nature of the postoperative evaluations (e.g., assessing sensory or motor blockade) may reveal the anaesthetic technique. To reduce potential bias, all assessors will follow standardised assessment protocols.
  Data analysts will remain blinded to the treatment allocation during the analysis phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anaesthesia (GA) (Experimental): Participants randomized to this arm will receive general anaesthesia during outpatient primary total knee or total hip arthroplasty. General anaesthesia is administered using total intravenous anaesthesia with short-acting agents, primarily propofol and remifentanil, delivered intravenously according to routine clinical practice. Perioperative care apart from the assigned anaesthetic technique follows standard clinical protocols at each study site.
  Interventions: Drug: General Anaesthesia
- Spinal Anaesthesia (SA) (Experimental): Participants randomized to this arm will receive spinal anaesthesia during outpatient primary total knee or total hip arthroplasty. Spinal anaesthesia is administered as a single-shot intrathecal injection of bupivacaine. Optional intrathecal opioid adjuncts and light intravenous sedation may be used at the discretion of the anaesthesiologist to ensure patient comfort. All other perioperative care follows standard clinical practice at each study site.
  Interventions: Drug: Spinal Anesthesia (bupivacaine)

INTERVENTIONS:
Drug: General Anaesthesia — General anaesthesia is administered using total intravenous anaesthesia with short-acting agents, primarily propofol and remifentanil. Anaesthesia is delivered intravenously using target-controlled or rate-controlled infusion systems according to routine clinical practice. Airway management and adjunct medications are provided as clinically indicated. The intervention is limited to the intraoperative period, and all other perioperative care follows standard clinical protocols at each study site.
  Other Names: Total Intravenous Anaesthesia; TIVA; Propofol-Remifentanil Anaesthesia
  Arms: General Anaesthesia (GA)
Drug: Spinal Anesthesia (bupivacaine) — Spinal anaesthesia is administered as a single-shot intrathecal injection of bupivacaine prior to surgery. Optional intrathecal opioid adjuncts, with fentanyl or sufentanil, may be used to enhance analgesia according to routine clinical practice. Light intravenous sedation may be provided if needed for patient comfort. The intervention is limited to the intraoperative period, and all other perioperative care follows standard clinical protocols at each study site.
  Other Names: Neuraxial Anaesthesia; Spinal Block; Intrathecal Anaesthesia
  Arms: Spinal Anaesthesia (SA)

SUMMARY:
Total knee arthroplasty (TKA) and total hip arthroplasty (THA) are common operations used to treat severe joint disease, most often caused by osteoarthritis. An increasing number of these procedures are now performed as outpatient surgery, meaning that patients can go home on the same day as the operation. This can be beneficial for both patients and healthcare systems, but it requires safe and efficient anaesthetic care.

Two different types of anaesthesia are commonly used for these operations: general anaesthesia (where the patient is asleep) and spinal anaesthesia (where the lower part of the body is numbed). Both methods are well established and widely used. Previous studies suggest that the choice of anaesthesia may affect how quickly patients recover, how comfortable they feel after surgery, and whether they can be safely discharged on the day of surgery. However, most existing studies are based on retrospective data, and there is limited randomized evidence comparing these anaesthetic techniques in the outpatient setting.

The GASPS trial is a multicentre, randomized, phase IV clinical study that compares general anaesthesia and spinal anaesthesia in adults undergoing outpatient primary total knee or hip arthroplasty. A total of 600 participants will be included and randomly assigned to receive one of the two anaesthetic methods on the day of surgery. All participants will receive standard surgical and perioperative care, and both anaesthetic techniques are part of routine clinical practice.

The main aim of the study is to investigate whether the type of anaesthesia influences the chance of successful same-day discharge, defined as going home on the day of surgery without needing to be readmitted within 48 hours. The study will also examine recovery time, pain, nausea and vomiting, use of pain medication, complications, patient-reported recovery and function, and healthcare costs. In addition, patient experiences of anaesthesia and postoperative recovery will be explored through interviews in a smaller group of participants.

Participants will be followed using questionnaires and medical records from the day of surgery up to 12 months after the operation. The results of this study are expected to provide clear and reliable information to help guide anaesthetic care for patients undergoing outpatient hip and knee replacement surgery.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) and total hip arthroplasty (THA) are among the most frequently performed elective surgical procedures and are highly effective treatments for advanced joint disease, most commonly osteoarthritis. Over the past decade, improvements in surgical techniques, perioperative care pathways, anaesthetic management, and postoperative rehabilitation have enabled an increasing proportion of these procedures to be performed as outpatient surgery, allowing patients to return home on the day of surgery. Outpatient arthroplasty has the potential to improve patient satisfaction, reduce hospital length of stay, lower healthcare costs, and decrease the risk of hospital-acquired complications. However, achieving safe and successful same-day discharge requires carefully optimized perioperative care.

Anaesthetic management is a central component of outpatient arthroplasty pathways. Both general anaesthesia (GA) and spinal anaesthesia (SA) are routinely used for TKA and THA, and both techniques are well established with extensive safety data. Neuraxial anaesthesia has traditionally been associated with reduced intraoperative blood loss and certain postoperative complications, and it is commonly recommended in clinical guidelines for hip and knee arthroplasty. In contrast, modern general anaesthesia using short-acting intravenous agents may offer advantages in the outpatient setting, including predictable onset and offset, rapid recovery of motor function, and reduced postoperative nausea and vomiting when volatile agents are avoided.

Despite widespread clinical use of both techniques, the optimal choice of anaesthesia for outpatient TKA and THA remains uncertain. Much of the existing evidence comparing GA and SA is derived from retrospective observational studies and registry-based analyses. These studies often include mixed inpatient and outpatient populations and are subject to confounding by indication, as patients receiving GA frequently differ from those receiving SA with respect to comorbidity, functional status, or anticipated surgical complexity. As a result, it is difficult to determine whether observed differences in outcomes are attributable to the anaesthetic technique itself or to underlying patient characteristics. Randomized clinical trials specifically designed to compare GA and SA in the outpatient arthroplasty setting are scarce.

The GASPS (General Anaesthesia vs Spinal Anaesthesia: Patient Outcomes and Success in Outpatient Primary Total Knee and Hip Arthroplasty) trial was designed to address this evidence gap. GASPS is a multicentre, randomized, phase IV clinical trial comparing GA and SA in adults undergoing outpatient primary TKA or THA. The overarching aim of the trial is to generate high-quality randomized evidence on whether the choice of anaesthetic technique influences the likelihood of successful same-day discharge and postoperative recovery in outpatient arthroplasty.

A total of 600 participants will be enrolled across multiple orthopaedic centres in Sweden. Eligible patients scheduled for outpatient primary TKA or THA are randomized on the day of surgery to receive either GA or SA. Randomization is performed using a stratified permuted block design, with stratification by type of surgery (knee or hip arthroplasty) and study site, to ensure balanced allocation across groups. Allocation concealment is maintained until shortly before surgery. Due to the nature of the interventions, blinding of patients and clinical staff is not feasible; however, data analysts remain blinded during analysis.

Both anaesthetic techniques are delivered according to standardized protocols that reflect contemporary routine clinical practice. General anaesthesia is provided using total intravenous anaesthesia with short-acting agents, primarily propofol and remifentanil, administered by trained anaesthesiologists. Spinal anaesthesia is administered as a single-shot intrathecal block with bupivacaine, with optional intrathecal opioid adjuncts and light sedation as clinically indicated. No experimental drugs or procedures are introduced, and all perioperative care apart from the assigned anaesthetic technique follows local standard practice.

The primary outcome of the trial is successful same-day discharge, defined as discharge from hospital on the day of surgery without readmission within 48 hours. This outcome was chosen as a clinically meaningful and patient-relevant measure of perioperative success in outpatient arthroplasty, integrating both recovery efficiency and short-term safety. Successful same-day discharge reflects the combined effects of anaesthetic technique, surgical care, postoperative recovery, and early complication rates.

Secondary outcomes are designed to capture multiple dimensions of perioperative and postoperative recovery. These include perioperative time metrics related to anaesthesia induction, surgery, and recovery; early postoperative outcomes such as pain, nausea and vomiting, opioid consumption, mobilisation, and adverse events; and patient-reported outcomes assessing quality of recovery, function, and health-related quality of life. Recovery is conceptualized as a multi-phase process, ranging from early recovery in the postoperative care unit to longer-term recovery at home. Validated instruments such as the Quality of Recovery-15 (QoR-15), Knee injury and Osteoarthritis Outcome Score (KOOS), Hip disability and Osteoarthritis Outcome Score (HOOS), and EQ-5D-5L are used to assess these domains over time.

In addition to quantitative outcomes, the GASPS trial incorporates a qualitative component to explore patient experiences of anaesthesia and postoperative recovery. Semi-structured interviews are conducted with a subset of participants several weeks after surgery. This mixed-methods approach allows for a deeper understanding of patient perceptions, expectations, and experiences that may not be fully captured by standardized questionnaires, and provides important contextual information to complement clinical and patient-reported outcome data.

Participants are followed from the day of surgery up to 12 months postoperatively using a combination of medical record review and patient-completed questionnaires. Safety monitoring focuses on adverse events occurring in the immediate perioperative period, while longer-term follow-up captures functional outcomes, quality of life, healthcare utilization, and productivity losses. A health economic evaluation is embedded within the trial to compare GA and SA in terms of costs and quality-adjusted life years, with the aim of informing resource-efficient anaesthetic strategies for outpatient arthroplasty.

By integrating randomized clinical data, patient-reported outcomes, qualitative insights, and health economic analyses, the GASPS trial aims to provide a evaluation of the role of anaesthetic technique in outpatient total knee and hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has given their written consent to participate in the trial.
2. Planned for primary TKA or THA.
3. Adults aged 18 to 80 years at time of written consent.
4. ASA (American Society of Anaesthesiologists) classification 1 or 2, or 3 without significant functional impairment.
5. Scheduled start of surgery before 13:00.
6. Ability to communicate in Swedish, ensuring understanding of informed consent and follow-up procedures.

Exclusion Criteria:

1. Indication for surgery other than degenerative or inflammatory joint diseases (e.g. fracture).
2. Body mass index (BMI) > 35 kg/m.
3. Preoperative opioid use exceeding 20 mg oral morphine equivalents daily.
4. Haemoglobin < 120 g/L (sample no older than 3 months).
5. Known bleeding disorders, including coagulopathies.
6. Known allergies to investigational anaesthetic drugs (e.g., bupivacaine, remifentanil, or propofol).
7. Neurological conditions with persistent motor or sensory deficits.
8. Localised infections at the spinal injection site.
9. Determined by the surgical or anaesthesia team to be unsuitable for trial participation and/or outpatient surgery.
10. Women of childbearing potential (i.e., those who are fertile, following menarche and until becoming post-menopausal, unless permanently sterile)

    1. Who are not willing to use a highly effective method of contraception judged by the investigator, from the time of signing the informed consent, OR
    2. Who has a positive pregnancy test at enrolment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful Same-Day Discharge | Day of surgery to 48 hours after discharge
  Successful same-day discharge is defined as discharge from the hospital on the day of surgery without readmission within 48 hours after discharge. Discharge readiness is assessed by the treating clinical team according to routine clinical criteria. Readmissions are identified through medical record review and patient follow-up.

SECONDARY OUTCOMES:
Time From Start of Anaesthesia to Start of Surgery | Day of surgery
  Elapsed time from initiation of anaesthesia to the start of surgical incision, recorded intraoperatively.
Time to Discharge From Post-Anaesthesia Care Unit (PACU) | From intervention to time of discharge from PACU
  Time from the start of surgery to discharge from the postoperative recovery unit (Phase II), based on predefined discharge criteria.
Time to Fulfilment of Hospital Discharge Criteria | During the hospital stay for surgery.
  Time from the start of surgery to fulfilment of predefined criteria for discharge from hospital (Phase III), assessed by the clinical care team.
Time to First Successful Mobilisation | During the hospital stay for surgery.
  Time from the start of surgery to first successful mobilisation, defined as the ability to walk with tolerable pain, and to ascend or descend stairs if applicable.
Opioid Consumption | Day of surgery to postoperative day 35
  Postoperative opioid use converted to oral morphine equivalents (OME), recorded during hospital stay and reported by patients after discharge.
Quality of Recovery (QoR-15) | Postoperative day 1 to postoperative day 35
  Patient-reported quality of postoperative recovery measured using the Quality of Recovery-15 (QoR-15) questionnaire.
Postoperative Pain | Day of surgery to postoperative day 35
  Postoperative pain assessed using the Numeric Rating Scale (NRS) during hospital stay for surgery.
Pain during recovery | Baseline and, postoperative day 1 to postoperative day 35
  Pain, measured with items 11 and 12 of QoR-15 questionnarie
Functional Outcome After Surgery | Baseline, 4 weeks, 6 months, and 12 months postoperatively
  Patient-reported functional outcomes assessed using the Knee injury and Osteoarthritis Outcome Score (KOOS) for knee arthroplasty and the Hip disability and Osteoarthritis Outcome Score (HOOS) for hip arthroplasty.
Adverse Events and Serious Adverse Events | Start of anaesthesia to postoperative day 3
  Incidence, severity, and frequency of adverse events and serious adverse events related to the perioperative period.
Predefined adverse outcomes | Day of surgery to 35 days postoperativly
  Incidence and frequency of predefined adverse outcomes.
Blood transfusions | During the hospital stay for surgery.
  Units of blood transfusesd
Patient Experiences of Anaesthesia and Recovery | 14 to 60 days after surgery
  Patient-reported experiences of anaesthesia and postoperative recovery explored through semi-structured qualitative interviews.
Cost-Effectiveness (Incremental Cost-Effectiveness Ratio) | Baseline to 12 months postoperatively
  Incremental cost-effectiveness ratios (ICERs) comparing general anaesthesia and spinal anaesthesia, calculated as differences in total costs divided by differences in quality-adjusted life years (QALYs) gained. QALYs are derived from EQ-5D-5L measurements.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: Ethical Principles for Medical Research Involving Human Participants. JAMA. 2025 Jan 7;333(1):71-74. doi: 10.1001/jama.2024.21972. PMID 39425955
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qual Res Psychol. januari 2006;3(2):77-101.
- [Background] Gibon E, Parvataneni HK, Prieto HA, Photos LL, Stone WZ, Gray CF. Outpatient total knee arthroplasty: is it economically feasible in the hospital setting? Arthroplast Today. 2020 Mar 13;6(2):231-235. doi: 10.1016/j.artd.2020.02.004. eCollection 2020 Jun. PMID 32577469
- [Background] Huang A, Ryu JJ, Dervin G. Cost savings of outpatient versus standard inpatient total knee arthroplasty. Can J Surg. 2017 Feb;60(1):57-62. doi: 10.1503/cjs.002516. PMID 28234591
- [Background] Churchill L, Pollock M, Lebedeva Y, Pasic N, Bryant D, Howard J, Lanting B, Laliberte Rudman D. Optimizing outpatient total hip arthroplasty: perspectives of key stakeholders. Can J Surg. 2018 Dec 1;61(6):370-376. doi: 10.1503/cjs.016117. PMID 30265638
- [Background] Kelly MP, Calkins TE, Culvern C, Kogan M, Della Valle CJ. Inpatient Versus Outpatient Hip and Knee Arthroplasty: Which Has Higher Patient Satisfaction? J Arthroplasty. 2018 Nov;33(11):3402-3406. doi: 10.1016/j.arth.2018.07.025. Epub 2018 Aug 1. PMID 30143333
- [Background] Gauthier-Kwan OY, Dobransky JS, Dervin GF. Quality of Recovery, Postdischarge Hospital Utilization, and 2-Year Functional Outcomes After an Outpatient Total Knee Arthroplasty Program. J Arthroplasty. 2018 Jul;33(7):2159-2164.e1. doi: 10.1016/j.arth.2018.01.058. Epub 2018 Feb 5. PMID 29506929
- [Background] Greimel F, Maderbacher G, Zeman F, Grifka J, Meissner W, Benditz A. No Clinical Difference Comparing General, Regional, and Combination Anesthesia in Hip Arthroplasty: A Multicenter Cohort-Study Regarding Perioperative Pain Management and Patient Satisfaction. J Arthroplasty. 2017 Nov;32(11):3429-3433. doi: 10.1016/j.arth.2017.05.038. Epub 2017 May 26. PMID 28641966
- [Background] Nilsson U, Jaensson M, Dahlberg K, Hugelius K. Postoperative Recovery After General and Regional Anesthesia in Patients Undergoing Day Surgery: A Mixed Methods Study. J Perianesth Nurs. 2019 Jun;34(3):517-528. doi: 10.1016/j.jopan.2018.08.003. Epub 2018 Nov 20. PMID 30470465
- [Background] Macfarlane AJ, Prasad GA, Chan VW, Brull R. Does regional anesthesia improve outcome after total knee arthroplasty? Clin Orthop Relat Res. 2009 Sep;467(9):2379-402. doi: 10.1007/s11999-008-0666-9. Epub 2009 Jan 7. PMID 19130163
- [Background] Nilsson U, Gruen R, Myles PS. Postoperative recovery: the importance of the team. Anaesthesia. 2020 Jan;75 Suppl 1:e158-e164. doi: 10.1111/anae.14869. PMID 31903575
- [Background] Allvin R, Berg K, Idvall E, Nilsson U. Postoperative recovery: a concept analysis. J Adv Nurs. 2007 Mar;57(5):552-8. doi: 10.1111/j.1365-2648.2006.04156.x. PMID 17284272
- [Background] Calkins TE, Johnson EP, Eason RR, Mihalko WM, Ford MC. Spinal Versus General Anesthesia for Outpatient Total Hip and Knee Arthroplasty in the Ambulatory Surgery Center: A Matched-Cohort Study. J Arthroplasty. 2024 Jun;39(6):1463-1467. doi: 10.1016/j.arth.2023.12.020. Epub 2023 Dec 15. PMID 38103803
- [Background] Keulen MHF, Asselberghs S, Boonen B, Hendrickx RPM, van Haaren EH, Schotanus MGM. Predictors of (Un)successful Same-Day Discharge in Selected Patients Following Outpatient Hip and Knee Arthroplasty. J Arthroplasty. 2020 Aug;35(8):1986-1992. doi: 10.1016/j.arth.2020.03.034. Epub 2020 Mar 27. PMID 32307291
- [Background] Gazendam AM, Tushinski D, Patel M, Bali K, Petruccelli D, Winemaker M, DeBeer J, Gillies L, Best K, Fife J, Wood TJ. Causes and predictors of failed same-day home discharge following primary hip and knee total joint arthroplasty: a Canadian perspective. Hip Int. 2023 Jul;33(4):576-582. doi: 10.1177/11207000221111101. Epub 2022 Jul 17. PMID 35848135
- [Background] Gong MF, McElroy MJ, Li WT, Finger LE, Shannon M, Gabrielli AS, Tisherman RF, O'Malley MJ, Klatt BA, Plate JF. Reasons and Risk Factors for Failed Same-Day Discharge After Total Joint Arthroplasty. J Arthroplasty. 2024 Jun;39(6):1468-1473. doi: 10.1016/j.arth.2023.11.032. Epub 2023 Nov 29. PMID 38040065
- [Background] Kendall MC, Cohen AD, Principe-Marrero S, Sidhom P, Apruzzese P, De Oliveira G. Spinal versus general anesthesia for patients undergoing outpatient total knee arthroplasty: a national propensity matched analysis of early postoperative outcomes. BMC Anesthesiol. 2021 Sep 15;21(1):226. doi: 10.1186/s12871-021-01442-2. PMID 34525959
- [Background] Klavas DM, Karim A, Lambert BS, Ferris MS, Delgado D, Incavo SJ. Does Total Intravenous Anesthesia With Short-acting Spinal Anesthetics in Primary Hip and Knee Arthroplasty Facilitate Early Hospital Discharge? J Am Acad Orthop Surg. 2018 May 15;26(10):e221-e229. doi: 10.5435/JAAOS-D-17-00474. PMID 29688961
- [Background] Mulroy MF, Larkin KL, Hodgson PS, Helman JD, Pollock JE, Liu SS. A comparison of spinal, epidural, and general anesthesia for outpatient knee arthroscopy. Anesth Analg. 2000 Oct;91(4):860-4. doi: 10.1097/00000539-200010000-00017. PMID 11004038
- [Background] Harsten A, Kehlet H, Ljung P, Toksvig-Larsen S. Total intravenous general anaesthesia vs. spinal anaesthesia for total hip arthroplasty: a randomised, controlled trial. Acta Anaesthesiol Scand. 2015 Mar;59(3):298-309. doi: 10.1111/aas.12456. Epub 2014 Dec 18. PMID 25522681
- [Background] Harsten A, Kehlet H, Toksvig-Larsen S. Recovery after total intravenous general anaesthesia or spinal anaesthesia for total knee arthroplasty: a randomized trial. Br J Anaesth. 2013 Sep;111(3):391-9. doi: 10.1093/bja/aet104. Epub 2013 Apr 11. PMID 23578860
- [Background] Memtsoudis SG, Sun X, Chiu YL, Stundner O, Liu SS, Banerjee S, Mazumdar M, Sharrock NE. Perioperative comparative effectiveness of anesthetic technique in orthopedic patients. Anesthesiology. 2013 May;118(5):1046-58. doi: 10.1097/ALN.0b013e318286061d. PMID 23612126
- [Background] Johnson RL, Kopp SL, Burkle CM, Duncan CM, Jacob AK, Erwin PJ, Murad MH, Mantilla CB. Neuraxial vs general anaesthesia for total hip and total knee arthroplasty: a systematic review of comparative-effectiveness research. Br J Anaesth. 2016 Feb;116(2):163-76. doi: 10.1093/bja/aev455. PMID 26787787
- [Background] Duque M, Schnetz MP, Yates AJ Jr, Monahan A, Whitehurst S, Mahajan A, Kaynar AM. Impact of Neuraxial Versus General Anesthesia on Discharge Destination in Patients Undergoing Primary Total Hip and Total Knee Replacement. Anesth Analg. 2021 Dec 1;133(6):1379-1386. doi: 10.1213/ANE.0000000000005156. PMID 34784324
- [Background] Yap E, Wei J, Webb C, Ng K, Behrends M. Neuraxial and general anesthesia for outpatient total joint arthroplasty result in similarly low rates of major perioperative complications: a multicentered cohort study. Reg Anesth Pain Med. 2022 May;47(5):294-300. doi: 10.1136/rapm-2021-103189. Epub 2022 Jan 6. PMID 34992150
- [Background] Owens PL, Barrett ML, Raetzman S, Maggard-Gibbons M, Steiner CA. Surgical site infections following ambulatory surgery procedures. JAMA. 2014 Feb 19;311(7):709-16. doi: 10.1001/jama.2014.4. PMID 24549551
- [Background] Pivot D, Hoch G, Astruc K, Lepelletier D, Lefebvre A, Lucet JC, Beaussier M, Philippe HJ, Vons C, Triboulet JP, Grandbastien B, Aho Glele LS. A systematic review of surgical site infections following day surgery: a frequentist and a Bayesian meta-analysis of prevalence. J Hosp Infect. 2019 Feb;101(2):196-209. doi: 10.1016/j.jhin.2018.07.035. Epub 2018 Jul 30. PMID 30071265
- [Background] Rullan PJ, Xu JR, Emara AK, Molloy RM, Krebs VE, Mont MA, Piuzzi NS. Major National Shifts to Outpatient Total Knee Arthroplasties in the United States: A 10-Year Trends Analysis of Procedure Volumes, Complications, and Healthcare Utilizations (2010 to 2020). J Arthroplasty. 2023 Jul;38(7):1209-1216.e5. doi: 10.1016/j.arth.2023.01.019. Epub 2023 Jan 21. PMID 36693513
- [Background] Aynardi M, Post Z, Ong A, Orozco F, Sukin DC. Outpatient surgery as a means of cost reduction in total hip arthroplasty: a case-control study. HSS J. 2014 Oct;10(3):252-5. doi: 10.1007/s11420-014-9401-0. Epub 2014 Jul 12. PMID 25264442
- [Background] W-Dahl A, Kärrholm J, Rogmark C, Johansson O, Ighani Arani P, Mohaddes M, m.fl. Årsrapport 2024 Svenska Ledprotesregistret [Internet]. Svenska Ledprotesregistret; 2024 aug [citerad 13 september 2024]. Tillgänglig vid: http://refdocs.registercentrum.se/10.18158/i_2vVZosV
- [Background] Lie SA, Engesaeter LB, Havelin LI, Gjessing HK, Vollset SE. Mortality after total hip replacement: 0-10-year follow-up of 39,543 patients in the Norwegian Arthroplasty Register. Acta Orthop Scand. 2000 Feb;71(1):19-27. doi: 10.1080/00016470052943838. PMID 10743987
- [Background] Ethgen O, Bruyere O, Richy F, Dardennes C, Reginster JY. Health-related quality of life in total hip and total knee arthroplasty. A qualitative and systematic review of the literature. J Bone Joint Surg Am. 2004 May;86(5):963-74. doi: 10.2106/00004623-200405000-00012. PMID 15118039
- [Background] Cross WW 3rd, Saleh KJ, Wilt TJ, Kane RL. Agreement about indications for total knee arthroplasty. Clin Orthop Relat Res. 2006 May;446:34-9. doi: 10.1097/01.blo.0000214436.49527.5e. PMID 16672869